CLINICAL TRIAL: NCT06628453
Title: Continuous Glucose Monitoring for Management of Type 2 Diabetes in Pregnancy
Brief Title: CGM for Management of Type 2 Diabetes in Pregnancy
Acronym: CGM2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Ashley N. Battarbee, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300013640; 1R01HD113612 (NIH)
Record Dates: First submitted 2024-09-25; First posted 2024-10-08 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Type 2 Diabetes Mellitus (T2DM); Pregnancy
Keywords: Diabetes; Pregnancy; CGM
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Continuous Glucose Monitoring (Experimental): Real-time continuous glucose monitoring
  Interventions: Device: CGM
- Self-Monitoring of Blood Glucose (No Intervention): Self-monitoring of blood glucose (standard of care)

INTERVENTIONS:
Device: CGM — Real-time continuous glucose monitoring
  Arms: Continuous Glucose Monitoring

SUMMARY:
The goal of this clinical trial is to learn if continuous glucose monitoring works better than self-monitoring of blood glucose (fingersticks) to treat type 2 diabetes in pregnancy. It will also learn about all risk factors (biologic, personal, social) for maternal and infant complications in type 2 diabetes pregnancies. The main questions it aims to answer are:

1. Does continuous glucose monitoring improve infant outcomes compared to self-monitoring of blood glucose?
2. Does continuous glucose monitoring improve maternal diabetes control and other maternal outcomes compared to self-monitoring of blood glucose?
3. What other factors increase the risk of maternal and infant complications?

Participants will:

1. Use continuous glucose monitoring or self-monitoring of blood glucose to monitor blood sugar control from enrollment until delivery
2. Have blood drawn at enrollment, 24 weeks, 34 weeks and delivery to measure hemoglobin A1c levels and store blood for future analysis
3. Complete surveys about social support, environmental stressors, diabetes distress and glucose monitoring satisfaction at research visits
4. Have umbilical cord blood collected at delivery for analysis

DETAILED DESCRIPTION:
We will conduct a multicenter, open-label randomized controlled trial of pregnant individuals with T2DM to test the effectiveness of CGM at improving maternal and neonatal outcomes, compared to SMBG. All pregnant women who have T2DM will be screened for eligibility. If a patient is eligible, the study will be explained to them and if they consent to participate, they will be randomized centrally in a 1:1 ratio to CGM or SMBG.

Participants randomized to CGM will receive a Dexcom G7 CGM and be instructed how to apply it, access the CGM data, and how to interpret and respond to trend arrows and alerts. Participants will replace the CGM device with a new sensor every 10 days for the entire pregnancy. Participants randomized to SMBG will be instructed to perform SMBG at least 4 times daily (fasting and 1-hour or 2-hours postprandial) and share their glucose data with their provider according to standard care. In order to collect comparable assessments of glycemic control between the groups, participants randomized to SMBG will wear a masked CGM for 10 days after randomization (Visit 1) and after Visits 2 (24 weeks) and Visit 3 (34 weeks). All participants will be provided a glucometer if they do not already have one and will have HbA1c and maternal serum collected at enrollment (6-22 weeks) and all study visits (24 weeks, 34 weeks, and delivery).

We will utilize ACOG and ADA recommendations for glycemic targets in pregnancy a standardized protocol with graduated goals for glycemic control to ensure consistency across arms and study sites. For pregnant individuals randomized to CGM, the target range will be 63-140mg/dL. For pregnant individuals randomized to SMBG, the targets will be fasting <95mg/dL, 1-hour postprandial less than 140mg/dL and 2-hour postprandial less than 120mg/dL. CGM reports and glucose logs will be reviewed at least every 1-2 weeks, and therapy adjustments (insulin, metformin, diet and/or lifestyle) will be recommended if less than 70% of glucose values are at target, regardless of the method of glucose monitoring. Additional therapy adjustments will be encouraged to achieve greater than 70% glucose values at target so long as there is not significant hypoglycemia (i.e. greater than 4%).

Telehealth visits may be utilized in addition to outpatient in person visits at the discretion of the provider, but should be used similarly for the CGM and SMBG groups. This protocol for glycemic management will be followed at all times including both at outpatient visits and during inpatient antepartum hospitalization. Intrapartum glycemic control, fetal testing and timing and route of delivery will be determined by the clinical provider in accordance with ACOG recommendations. After birth, umbilical cord blood will be collected for metabolic analyses, and neonates will have a heelstick performed to measure capillary blood glucose as part of usual care given maternal T2DM. Additional care including NICU admission and treatment of hypoglycemia will be at the discretion of the neonatal provider.

Validated screening tools to assess different SDoH domains will be administered at the first 2 study visits. At enrollment, each participant will be administered the Protocol for Responding to and Assessing Patient Assets, Risks and Experiences (PRAPARE) survey, a validated screening tool designed to identify SDoH including personal factors, family and housing, money and resources, and social and emotional health and safety. The home address provided will be used to calculate SVI and area deprivation index (ADI), a measure created to assess socioeconomic disadvantage at a neighborhood level based on income, education, employment and housing quality. Participants will complete the U.S. Adult Household Food Security Survey Module (HFSSM), a 10-item self-report questionnaire aimed at assessing food security over the prior 12 months as food insecurity may be associated with adverse outcomes. Participants will also complete the Type 2 Diabetes Distress Assessment System (T2-DDAS), a 29-item survey designed to identify the overall amount of DM-related distress as well as the sources of stress including hypoglycemia, long-term health, healthcare provider, interpersonal issues, shame or stigma, healthcare access, and management demands. At visit 2, participants will complete the Short Assessment of Health Literacy (SAHL) and the Diabetes Numeracy Test 15 (DNT15) given association between lower educational attainment and health literacy and numeracy with worse outcomes. Participants will also complete the Multidimensional Scale of Perceived Social Support (MSPSS), the only self-reported measure in a study of psychosocial stress associated with adverse pregnancy outcomes and the Experiences of Discrimination (EOD) scale, a 9-item self-report about lifetime experiences of discrimination attributed to race, ethnicity or skin color. At delivery, participants will repeat the T2-DDAS to assess if CGM impacted DM distress and complete a Glucose Monitoring Satisfaction Survey (GMSS), a validated tool to assess satisfaction with the assigned method of glucose monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus treated with daily insulin injections or oral hypoglycemic agents diagnosed before pregnancy or at less than 14 weeks gestation with hemoglobin A1c 6.5% or greater
* Pregnant with viable fetus at 6 to less than 23 weeks gestation
* Maternal age 18-50 years old

Exclusion Criteria:

* Unable or unwilling to wear CGM due to intolerance to medical-grade adhesives or skin conditions
* Multiple gestation
* Major fetal anomaly or two or more minor fetal anomalies
* Planned delivery outside study consortium
* Participating in another conflicting interventional study
* Participation in this trial in a previous pregnancy
* Patient unable to consent
* Physician refusal for other reasons

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 564 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Time in Range (TIR) at 34 weeks gestation | 33 to 35 weeks gestation
  Percentage of time spent within target range (63-140mg/dL) on Continuous Glucose Monitoring at 34 weeks gestation
Composite Neonatal Morbidity | From the date of delivery to the date of neonatal hospital discharge, assessed up to 12 months of life
  Composite morbidity of the neonate including one or more of preterm birth (delivery less than 37 weeks for any indication), birth trauma (shoulder dystocia with nerve injury, clavicular or humeral fracture or 3 or more maneuvers to resolve), hypoglycemia (requiring treatment with dextrose gel or IV within 24 hours of birth), hyperbilirubinemia (requiring phototherapy within 72 hours of birth), large-for-gestational-age infant (birthweight greater than the 90th percentile for gestational age), and miscarriage, stillbirth or neonatal death prior to hospital discharge.

SECONDARY OUTCOMES:
Preterm birth | Delivery
  Delivery less than 37 weeks gestation
Birth trauma | Delivery
  Shoulder dystocia with nerve injury, clavicular or humeral fracture or 3 or more maneuvers to relieve
Neonatal hypoglycemia | Delivery to 24 hours of life
  Low neonatal glucose requiring treatment with dextrose gel or IV within 24 hours of life
Hyperbilirubinemia | Delivery to 72 hours of life
  Elevated bilirubin requiring phototherapy within 72 hours of life
Large-for-gestational-age (LGA) neonate | Delivery
  Birthweight greater than the 90th percentile for gestational age
Small-for-gestational-age (SGA) neonate | Delivery
  Birthweight less than the 10th percentile for gestational age
Fetal glucose | Delivery
  Concentration of umbilical cord blood glucose (mg/dL)
Fetal insulin | Delivery
  Concentration of umbilical cord blood insulin (uU/mL)
Fetal C-peptide | Delivery
  Concentration of umbilical cord blood C-peptide (ng/mL)
Fetal leptin | Delivery
  Concentration of umbilical cord blood leptin (ng/mL)
Fetal ghrelin | Delivery
  Concentration of umbilical cord blood ghrelin (uU/L)
Fetal surfactant protein D | Delivery
  Concentration of umbilical cord blood surfactant protein D (ng/mL)
Time Above Range (TAR) at 34 weeks | 33 to 35 weeks
  Percentage of time spent above range greater than 140mg/dL on Continuous Glucose Monitoring (CGM) at 34 weeks
Time Below Range (TBR) at 34 weeks | 33 to 35 weeks
  Percentage of time spent below range less than 63mg/dL on Continuous Glucose Monitoring at 34 weeks
Mean glucose at 34 weeks | 33 to 35 weeks
  Average glucose in mg/dL using Continuous Glucose Monitoring data at 34 weeks
Glucose Management Indicator (GMI) | 33 to 35 weeks
  Glucose management indicator as an estimate of hemoglobin A1c calculated using mean glucose on CGM at 34 weeks
Glucose variability at 34 weeks | 33 to 35 weeks
  Coefficient of variation calculated as the mean glucose divided by standard deviation using Continuous Glucose Monitoring data at 34 weeks
Mean fasting glucose at 34 weeks | 33 to 35 weeks
  Average glucose at 6-7am on Continuous Glucose Monitoring at 34 weeks
Hemoglobin A1c at Delivery | Delivery
  Hemoglobin A1c (%) at delivery
Insulin total daily dose at delivery | Delivery
  Total number of units of insulin taken per day at time of delivery
Cesarean delivery | Delivery
  First cesarean delivery or cesarean delivery after a history of prior cesarean
Glucose Monitoring Satisfaction | Delivery
  Score on glucose monitoring satisfaction survey at delivery
Fetal or neonatal death | From the date of randomization to the date of neonatal hospital discharge, assessed up to 12 months of life
  Miscarriage (pregnancy loss less than 20 weeks), stillbirth (fetal death at 20 weeks or more), or neonatal death (death after birth up to 28 days of life)
Neonatal Intensive Care Unit (NICU) Admission | From the date of delivery to the date of neonatal hospital discharge, assessed up to 12 months of life
  Admission to the neonatal intensive care unit with length of stay greater than 24 hours
Neonatal length of stay | From the date of delivery to the date of neonatal hospital discharge, assessed up to 12 months of life
  Duration of neonatal hospitalization after delivery
Neonatal mechanical ventilation | From the date of delivery to the date of neonatal hospital discharge, assessed up to 12 months of life
  Neonate requiring intubation and mechanical ventilation for respiratory support
Insulin increase during pregnancy | From the date of randomization to the date of delivery, assessed up to 9 months
  Percentage change in total daily dose of insulin at delivery compared to enrollment
Preeclampsia | From the date of randomization to the date of maternal hospital discharge after delivery, assessed up to 9 months
  Elevated blood pressure greater than 140/90 mmHg after 20 weeks gestation with proteinuria or other severe features by ACOG criteria (may be superimposed on chronic hypertension or not)
Postpartum infection | From the date of delivery through 6 weeks' postpartum
  Developing one or more of endometritis, wound infection or other wound complication such as seroma, hematoma or dehiscence)
Glucose Monitoring Adherence | From the date of randomization to the date of delivery, assessed up to 9 months
  Defined as percentage of expected self-monitoring of blood glucose (SMBG) values completed based on recommended 4 values per day for participants in the SMBG arm and percentage of time Continuous Glucose Monitoring (CGM) in use in the CGM arm

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Battarbee, MD, MSCR, Principal Investigator — University of Alabama at Birmingham
Locations (7):
- United States (7):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California at San Diego, San Diego, California
  - University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - University of Texas Health Science Center at Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
All data produced in the course of the project will be preserved and shared including:
  1. Recruitment rates, reasons for refusal, adherence, loss to follow up
  2. Demographics and clinical data
  3. Glucose and laboratory values
  4. Satisfaction and survey responses
Supporting Information: Study Protocol
Time Frame: Data will be made available at the time of publication or the end of the funding period, whichever comes first.
Access Criteria: Deidentified individual patient data will be deposited in the NICHD DASH repository with public access. There is no planned requirement for data use agreements at this time; however, we will monitor the sensitive nature of study data collected at each of the participating sites and revise if needed during the conduct of the trial.

REFERENCES:
- [Background] Padgett CE, Ye Y, Champion ML, Fleenor RE, Orfanakos VB, Casey BM, Battarbee AN. Continuous Glucose Monitoring for Management of Type 2 Diabetes and Perinatal Outcomes. Obstet Gynecol. 2024 Nov 1;144(5):677-683. doi: 10.1097/AOG.0000000000005609. Epub 2024 May 23. PMID 38781595